CLINICAL TRIAL: NCT02785705
Title: Immunogenicity and Safety Evaluation of Bivalent Types 1 and 3 Oral Poliovirus Vaccine by Comparing Different Poliomyelitis Vaccination Schedules in Chinese Infant: a Randomized Controlled Non-Inferiority Clinical Trial
Brief Title: Randomized Controlled Trial for Immunogenicity and Safety Evaluation of Bivalent Types 1 and 3 Oral Poliovirus Vaccine
Acronym: TTbOPV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guangxi Zhuang Autonomous Region Center for Disease Prevention and Control (Other Government)
Collaborators: Air Force Military Medical University, China (Other); Beijing Tiantan Biological Products Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zhaojun Mo, Director, Guangxi Zhuang Autonomous Region Center for Disease Prevention and Control
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Tiantan-201417903
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Poliomyelitis
Keywords: immunization; vaccine schedule; poliomyelitis; polio; oral polio vaccine; inactivated polio vaccine
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- cIPV-bOPV-bOPV poliovirus vaccine (Experimental): Participants would be vaccine with trivalent conventional inactivated poliovirus vaccine, and two bivalent types 1 and 3 oral poliovirus vaccine sequentially.
  Interventions: Biological: poliovirus vaccine
- cIPV-tOPV-tOPV poliovirus vaccine (Experimental): Participants would be vaccine with trivalent conventional inactivated poliovirus vaccine, and two trivalent types 1, 2 and 3 oral poliovirus vaccine sequentially.
  Interventions: Biological: poliovirus vaccine
- cIPV-cIPV-bOPV poliovirus vaccine (Experimental): Participants would be vaccine with two shots of trivalent conventional inactivated poliovirus vaccine, and one bivalent types 1 and 3 oral poliovirus vaccine sequentially.
  Interventions: Biological: poliovirus vaccine
- cIPV-cIPV-tOPV poliovirus vaccine (Experimental): Participants would be vaccine with two shots of trivalent conventional inactivated poliovirus vaccine, and one trivalent types 1, 2 and 3 oral poliovirus vaccine sequentially.
  Interventions: Biological: poliovirus vaccine
- cIPV-cIPV-cIPV poliovirus vaccine (Experimental): Participants would be vaccine with three shots of trivalent conventional inactivated poliovirus vaccine.
  Interventions: Biological: poliovirus vaccine
- tOPV-tOPV-tOPV poliovirus vaccine (Experimental): Participants would be vaccine with three times of trivalent types 1, 2 and 3 oral poliovirus vaccine .
  Interventions: Biological: poliovirus vaccine

INTERVENTIONS:
Biological: poliovirus vaccine — Different vaccination schedules with bOPV, tOPV and cIPV would be provided for 6 arms respectively.
  Other Names: bivalent types 1 and 3 oral poliovirus vaccine; trivalent conventional inactivated poliovirus vaccine; trivalent types 1, 2 and 3 oral poliovirus vaccine

SUMMARY:
Type 2 component of oral poliovirus vaccine is slated for global withdrawal through a switch from trivalent oral poliovirus vaccine (tOPV) to bivalent oral poliovirus vaccine (bOPV) for preventing paralytic polio caused by circulating vaccine-derived poliovirus type 2. We aimed to assess immunogenicity and safety profile of six vaccination schedules with different sequential doses of inactivated poliovirus vaccine (IPV), tOPV, or bOPV.

DETAILED DESCRIPTION:
A randomized controlled trial was conducted in China in 2015. After informed consent was obtained from a parent or legally acceptable representative, healthy newborn babies were randomly allocated to one of six groups: cIPV-bOPV-bOPV, cIPV-tOPV-tOPV, cIPV-cIPV-bOPV, cIPV-cIPV-tOPV, cIPV-cIPV-cIPV, and tOPV-tOPV-tOPV. The key eligibility criteria were: full-term birth (37-42 weeks of gestation), birthweight ≥2·5 kg, no obvious medical disorders and no polio vaccination. Infants received following three doses sequentially with 4- 6 weeks interval after collecting blood sample: cIPV-bOPV-bOPV, cIPV-tOPV-tOPV, cIPV-cIPV-bOPV, cIPV-cIPV-tOPV, cIPV-cIPV-cIPV, and tOPV-tOPV-tOPV; and will be proactively followed up for observing adverse events after the first dose and 30 days after all doses. Antibodies of type 1, 2, and 3 poliovirus were tested 30 days after the third dose. The primary study objective was to investigate immunogenicity and safety profile of different vaccine schedules, evaluated by seroconversion, seroprotection and antibody titre against poliovirus types 1, 2, and 3 in the per-protocol population.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were healthy full-term (37-42 weeks) infants aged 60-90 days who weighed more than 2·5 kg at birth with no obvious medical disorders, no polio vaccination, no immunoglobulin vaccinated, no other attenuated vaccine immured in the past 14 days and no other inactivated vaccine immured.

Exclusion Criteria:

* Participants were excluded if meet one or more of following criteria: were or were at risk of immunodeficiency, severe allergic reaction, acute fever and infectious diseases, severe chronic diseases, family history of allergies, convulsions, seizures, encephalopathy and psychiatric diseases, oral steroids at least 14 consecutive days in the past month, axillary temperature equal or greater than 38·0°C in the past three days, diarrhea (defection frequency equal or greater than three times per day) in the past seven days, and participated in other drug clinical trials.

Ages: 60 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Proportion of infants with seroconversion | 30 days after vaccination
  Primary immunogenicity outcome was the proportion of infants with seroconversion, which was defined as the 30 days post-vaccination titer equal or greater than eight for susceptible infants and the post-vaccination titer is four times higher than pre-vaccination titer for unsusceptible infants. Here, susceptible infants are the ones whose pre-vaccination titer less than eight. Otherwise, the subjects are categories as unsusceptible ones.

SECONDARY OUTCOMES:
Overall seroprotection rate | 30 days after vaccination
  Overall seroprotection rate was defined as the proportion of subjects with reciprocal titre of at least eight.
Geometric mean of antibody titres (GMT) | 30 days after vaccination
Increase of geometric mean of antibody titres (GMI) | 30 days after vaccination
Proportion of infants with serious adverse events | Six months after vaccination
Solicited adverse events | 30 days after vaccination
  Solicited adverse events involving both systemic reactions (including fever, irritability/fussiness, somnolence, vomit, diarrhea, and allergic reaction) and local reactions (including tenderness, redness, swelling, and callous around the injection sites).

OTHER OUTCOMES:
Proportion of infants with seroconversion in susceptible population | 30 days after vaccination
  Proportion of infants with seroconversion, which was defined as the 30 days post-vaccination titer equal or greater than eight for susceptible infants. Here, susceptible infants are the ones whose pre-vaccination titer less than eight.
Proportion of infants with seroconversion in unsusceptible population | 30 days after vaccination
  Proportion of infants with seroconversion, which was defined as the 30 days post-vaccination titer is four times higher than pre-vaccination titer for unsusceptible infants.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaojun Mo, Principal Investigator — Center of Diseases Control and Prevention (CDC) of Hezhou County and Zhongshan County in Guangxi Zhuang Autonomous Region in China

IPD SHARING:
Plan to Share IPD: No